CLINICAL TRIAL: NCT05306119
Title: Developing a Method of Rehabilitation for Patients After Myocardial Revascularization Combined With Low Back Pain and Criteria for Evaluating Its Effectiveness
Brief Title: Developing a Method of Rehabilitation for Patients After Myocardial Revascularization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gomel State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20213753
Record Dates: First submitted 2022-01-06; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-01

CONDITIONS: Rehabilitation; Low Back Pain; Revascularization
Keywords: Rehabilitation; Revascularization; Low back pain; myocardial revascularization
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Main group (Active Comparator): Patients with low back pain who had undergone myocardial revascularization surgery within a year prior to admission to a sanatorium organization, admitted for a course of sanatorium treatment with an individual program of medical rehabilitation with the use of means, affecting both diseases lasting up to 21 days
  Interventions: Other: Rehabilitation method
- Comparison group (No Intervention): Patients with low back pain who had undergone myocardial revascularization surgery within a year prior to admission to a sanatorium organization, admitted for a course of sanatorium treatment lasting up to 21 days
- Control group (No Intervention): Healthy people aged 40-60 y.o.

INTERVENTIONS:
Other: Rehabilitation method — Application of techniques of kinesiotherapy, electrotherapy, massage in comorbid patients and patients with low back pain who had undergone myocardial revascularization surgery in main group.
  Arms: Main group

SUMMARY:
As a result, will be developed:

a list of criteria for functional impairment in patients after myocardial revascularization combined with low back pain; a list of criteria for disabilities in patients after myocardial revascularization combined with low back pain; method of medical rehabilitation of patients after myocardial revascularization combined with low back pain; and criteria for evaluating its effectiveness.

DETAILED DESCRIPTION:
Aim: to improve the quality of medical rehabilitation of patients after myocardial revascularization combined with low back pain by developing the method of medical rehabilitation with evaluating its effectiveness.

Objectives:

1. To exam clinical and functional state assessment of patients after myocardial revascularization combined with low back pain.
2. To analyze functional status of patients after myocardial revascularization combined with low back pain, who were admitted for medical rehabilitation and determine a list of criteria of impaired functions and a list of criteria for life limitation in patients after myocardial revascularization combined with low back pain.
3. To develop an algorithm for assessing patients' functional status after myocardial revascularization combined with low back pain.
4. To analyze of the effect of different means and methods of rehabilitation in comorbid patients after myocardial revascularization combined with low back pain: the degree of severity of pain syndrome, limitation of mobility, ability to self-care.
5. To develop the Draft Electronic Medical Rehabilitation Card of a patient (a medical rehabilitation card of a standard pattern).
6. Choose the most effective techniques of medical rehabilitation, determining the efficiency of performed of medical rehabilitation measures in patients after myocardial revascularization combined with low back pain and form a list of medical rehabilitation measures in these patients.
7. To evaluate the effectiveness of medical rehabilitation in patients after myocardial revascularization combined with low back pain and list of them.
8. To develop a method of medical rehabilitation of patients after myocardial revascularization combined with low back pain.
9. Evaluate the effectiveness of the developed method of medical rehabilitation of patients after myocardial revascularization combined with low back pain in the medium term (in the period of 6 months, 1 year after the end of rehabilitation).
10. To evaluate the effectiveness of medical rehabilitation of patients after myocardial revascularization combined with low back pain and approve the developed indicators in order to evaluate the efficiency of medical rehabilitation in this group of patients.
11. To develop an instruction manual containing a method of medical rehabilitation in patients after myocardial revascularization combined with low back pain and criteria for assessing its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Patients After Myocardial Revascularization Combined With Low Back Pain of 40-60 years of age

Exclusion Criteria:

* Arterial hypertension
* Heart attack
* Atherosclerosis
* Stroke
* Coronary heart disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Back pain | 21 days after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Heartache | 21 days after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Angina pectoris | 21 days after intervention of rehabilitation method
  ECG. Reveal the signs of ischemia (deviation of ST segment).
Arrhythmia | 21 days after intervention of rehabilitation method
  Holter monitor. Assessment of painless ischemia, heart rhythm disorders, silent ischemia.
Exercise tolerance | 21 days after intervention of rehabilitation method
  Treadmill Exercise Stress Test. Assessment of exercise tolerance, coronary reserve.
Paresis | 21 days after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Blood pressure level | 21 days after intervention of rehabilitation method
  Systolic blood pressure and Diastolic blood pressure is measured in units of millimeters of mercury (mmHg)
Mobility | 21 days after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Self-service | 21 days after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Work capacity | 21 days after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Back pain | 6 months after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Heartache | 6 months after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Angina pectoris | 6 months after intervention of rehabilitation method
  ECG. ECG. Reveal the signs of ischemia (deviation of ST segment).
Arrhythmia | 6 months after intervention of rehabilitation method
  Holter monitor. Assessment of painless ischemia, heart rhythm disorders, silent ischemia.
Exercise tolerance | 6 months after intervention of rehabilitation method
  Treadmill Exercise Stress Test. Assessment of exercise tolerance, coronary reserve.
Paresis | 6 months after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Blood pressure level | 6 months after intervention of rehabilitation method
  Systolic blood pressure and Diastolic blood pressure is measured in units of millimeters of mercury (mmHg)
Mobility | 6 months after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Self-service | 6 months after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Work capacity | 6 months after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Back pain | 1 year after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Heartache | 1 year after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Angina pectoris | 1 year after intervention of rehabilitation method
  ECG. Reveal the signs of ischemia (deviation of ST segment).
Arrhythmia | 1 year after intervention of rehabilitation method
  Holter monitor. Assessment of painless ischemia, heart rhythm disorders, silent ischemia.
Exercise tolerance | 1 year after intervention of rehabilitation method
  Treadmill Exercise Stress Test. Assessment of exercise tolerance, coronary reserve.
Paresis | 1 year after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Blood pressure level | 1 year after intervention of rehabilitation method
  Systolic blood pressure and Diastolic blood pressure is measured in units of millimeters of mercury (mmHg)
Mobility | 1 year after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance
Self-service | 1 year after intervention of rehabilitation method
  Self-report according to the questionnaire Short Form Medical Outcomes Study SF-36. (SF-36, 1998), ranges from 0 to 100.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Work capacity | 1 year after intervention of rehabilitation method
  Visual examination with a determination of a degree
  The Oxford Scale
  The most commonly accepted method of evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  Flicker of movement Through full range actively with gravity counterbalanced Through full range actively against gravity Through full range actively against some resistance Through full range actively against strong resistance

SECONDARY OUTCOMES:
Stroke | 21 days after intervention of rehabilitation method
  SCORE 2 chart Risk assessment of cardiovascular accidents. A scale for assessing the risk of death due to cardiovascular disease within 10 years. Assessment is based on the age, sex, systolic pressure (mm.Hg), cholesterol level (mmol/l), smoking status.
  Scores: < 1%, 1%, 2 %, 3-4 %, 5-9 %, 10-14 %, 15% and over.
Acute myocardial infarction | 21 days after intervention of rehabilitation method
  Increasing levels of cardiac specific biomarkers (CK-MB, Myoglobin, Troponin T and I), ECG, Echocardiography, SCORE 2021 chart, pain (self-report).
Death due to vascular diseases | 21 days after intervention of rehabilitation method
  The Lown grading system for ventricular arrhythmias of high rank The Lown grading system is used in observational and experimental studies of ischaemic heart disease. This grading system uses three levels of ventricular premature depolarisation frequency and four complex features to assign patients to one of seven grades.
  Assessment occurs depending on the number and type of extrasystoles according to Holter monitoring data.
  Grades: 0, 1, 2, 3A, 3B, 4A, 4B, 5.
Stroke | 6 months after intervention of rehabilitation method
  SCORE 2 chart Risk assessment of cardiovascular accidents. A scale for assessing the risk of death due to cardiovascular disease within 10 years. Assessment is based on the age, sex, systolic pressure (mm.Hg), cholesterol level (mmol/l), smoking status.
  Scores: < 1%, 1%, 2 %, 3-4 %, 5-9 %, 10-14 %, 15% and over.
Acute myocardial infarction | 6 months after intervention of rehabilitation method
  Increasing levels of cardiac specific biomarkers (CK-MB, Myoglobin, Troponin T and I), ECG, Echocardiography, SCORE 2021 chart, pain (self-report).
Death due to vascular diseases | 6 months after intervention of rehabilitation method
  The Lown grading system for ventricular arrhythmias of high rank The Lown grading system is used in observational and experimental studies of ischaemic heart disease. This grading system uses three levels of ventricular premature depolarisation frequency and four complex features to assign patients to one of seven grades.
  Assessment occurs depending on the number and type of extrasystoles according to Holter monitoring data.
  Grades: 0, 1, 2, 3A, 3B, 4A, 4B, 5.
Stroke | 1 year after intervention of rehabilitation method
  SCORE 2 chart Risk assessment of cardiovascular accidents. A scale for assessing the risk of death due to cardiovascular disease within 10 years. Assessment is based on the age, sex, systolic pressure (mm.Hg), cholesterol level (mmol/l), smoking status.
  Scores: < 1%, 1%, 2 %, 3-4 %, 5-9 %, 10-14 %, 15% and over.
Acute myocardial infarction | 1 year after intervention of rehabilitation method
  Increasing levels of cardiac specific biomarkers (CK-MB, Myoglobin, Troponin T and I), ECG, Echocardiography, SCORE 2021 chart, pain (self-report).
Death due to vascular diseases | 1 year after intervention of rehabilitation method
  The Lown grading system for ventricular arrhythmias of high rank The Lown grading system is used in observational and experimental studies of ischaemic heart disease. This grading system uses three levels of ventricular premature depolarisation frequency and four complex features to assign patients to one of seven grades.
  Assessment occurs depending on the number and type of extrasystoles according to Holter monitoring data.
  Grades: 0, 1, 2, 3A, 3B, 4A, 4B, 5.

CONTACTS AND LOCATIONS:
Overall Officials: Natalliya Halinouskaya, Proff, Study Director — Gomel State Medical University
Locations (1):
- Gomel State Medical University, Homyel, Province, Belarus

IPD SHARING:
Plan to Share IPD: No